CLINICAL TRIAL: NCT06151223
Title: A Prospective Registry for Patients at High-Risk for Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-012752
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; PDAC; PDAC - Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — All samples will be stored for future analysis in the Molecular Cancer Diagnostic Laboratory and Biospecimens Accessioning and Processing (BAP) at Mayo Clinic. All biospecimens will be stored in a bar-coded manner with unique study IDs. No permanent cell lines be established. This study involves testing of methylated DNA for research purposes only. Future studies may include whole genome sequencing. This information will not be documented in the subject's medical record and subjects will not be notified of results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tier 1: * Participants with Peutz-Jeghers syndrome and/or carriers of a germline CDKN2A mutation and/or hereditary pancreatitis with PRSS1 mutation and clinical history of pancreatitis(age ≥40 or 10 years younger than youngest affected blood relative)
  * Carriers of a germline BRCA2, BRCA1, PALB2, ATM, MLH1, MSH2, or MSH6 gene mutation with at least one affected first-degree blood relative (age ≥45 or 10 years younger than youngest affected blood relative)
  * At least one first-degree relative (FDR) with pancreatic cancer who in turn also has a first-degree relative with pancreatic cancer and/or at least two affected blood relatives on the same side of the family, of whom at least one is an FDR to the individual and/or at least three affected relatives on the same side of the family, of whom at least one is an FDR to the individual(age ≥50 or 10 years younger than youngest affected blood relative)
  Interventions: Other: Bio-specimen Collection: Blood; Other: Bio-specimen Collection: Pancreatic Juice
- Tier 2: * Individual with family history of PDAC in only one first degree relative (FDR); age ≥50 or 10 years younger than the affected first degree relative
  * OR known BRCA2, BRCA1, PALB2, ATM, MLH1, MSH2, or MSH6 gene mutation; age > 45 who do not meet tier 1 criteria.
  Interventions: Other: Bio-specimen Collection: Blood; Other: Bio-specimen Collection: Pancreatic Juice; Diagnostic Test: MRI

INTERVENTIONS:
Other: Bio-specimen Collection: Blood — At study enrollment and prior to any pancreatic surgery and prior to or at least 3 days after the most recent GI endoscopy procedure, approximately 50 ml (10 teaspoons) of blood will be drawn from all participants and be processed according to standardized study biospecimen protocol. Serial blood collection will be offered to all the participants depending on the subjects' tier classification. Blood draw will be completed at Mayo Clinic when the subjects come back, or study blood draw kit may be sent for external collection.
  Other Names: Blood Draw
Other: Bio-specimen Collection: Pancreatic Juice — This may be collected from research subjects every time they are undergoing a clinically indicated endoscopic ultrasound (EUS), endoscopic retrograde cholangiopancreatography (ERCP) or upper gastrointestinal endoscopy (EGD) procedure. Pancreatic juice will not be collected if PI or provider determines it is not in the best interest of the subject. Pancreatic juice collection will be performed prior to fine needle aspiration (FNA), brushing or stent placements if performed during the same endoscopic procedure.
  Other Names: Pancreatic Juice Collection
Diagnostic Test: MRI — A research MRI with contrast that includes a Magnetic Resonance Cholangiopancreatography (MRCP) will be offered to patients in the Tier 2 cohort at baseline and at 3-year intervals if not done as standard of care. Gadolinium based intravascular contrast will be administered for this procedure. Sedation for claustrophobia/anxiety per clinical protocol will be an option if the patients requested. Subject would be notified of any concerning results. A safety questionnaire will be completed by the study team before ordering the MRI.
  Clinically indicated MRIs for the TIER 1 participants will be used and collected as part of the registry.
  If a clinical MRI/MRCP has been performed between 0 to 3 months before obtaining consent, the prior clinical MRI/MRCP could be used to obtain baseline imaging data.
  Other Names: Magnetic Resonance Imaging
  Groups: Tier 2

SUMMARY:
This study aims to facilitate discovery and validation of tests for early detection in subjects at high risk for pancreatic ductal adenocarcinoma (PDAC) and to facilitate the use of state-of-the-art machine learning-based algorithms that utilize databases and images with the purpose of identifying early stages of pancreatic cancer, as well as people at high-risk.The study also aims to provide a platform for development of an interventional protocol for early detection of PDAC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Able to provide written informed consent
* Meets criteria as a High-Risk Individual as defined by protocol

Exclusion Criteria:

* Individual who has a personal history of pancreatic ductal adenocarcinoma (PDAC)
* History of total pancreatectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants at high risk of PDAC will be identified from the providers' calendars, provider referrals, and Mayo Clinic databases.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2031-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Collection of biospecimen samples (blood and pancreatic juice) | Up to 10 years
  Sufficient biospecimens (blood and pancreatic juice) will be collected in 10 years from participants to provide a resource for nested case-control studies of promising biomarkers for discovery and validation of tests for early detection in subjects at high risk for pancreatic ductal adenocarcinoma (PDAC)..
Collection of radiology images and videos | Up to 10 years
  Collect and archive radiology images and videos obtained during esophagogastroduodenoscopy (EDG)-endoscopic ultrasound (EUS) and endoscopic retrograde cholangiopancreatography (ERCP) in high risk individuals undergoing screening and surveillance tests. An imaging dataset designed for studies of promising imaging biomarkers and developing AI-assisted algorithms can be collected within10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Shounak Majumder, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials